CLINICAL TRIAL: NCT05246189
Title: Employment Retention Issues for Patient With Pseudoxanthoma Elasticum
Brief Title: Employment of Patients With Pseudoxanthoma Elasticum
Acronym: MEE-PXE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A03008-33
Record Dates: First submitted 2022-01-21; First posted 2022-02-18 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-02

CONDITIONS: Pseudoxanthoma Elasticum; Employment
Keywords: Employment retention; DIsease impact
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with PXE working aged: Patient diagnosed with PXE on working age and followed up by the French Reference Center.
  Interventions: Other: Telephone Call

INTERVENTIONS:
Other: Telephone Call — Eligible subjects will be pre-selected by the study investigators on the basis of the medical file. A letter of information about the study will be sent to all the pre-selected eligible patients, with the exception of patients who have expressed an objection to the processing of their data for research purposes during their treatment.
  The investigators will contact eligible patients by telephone approximately 2 weeks after the mailing of the information letter. During this telephone call, the investigator will answer any questions the patient may have about the study and will collect the patient's non-objection to participate in the study and their responses to the questionnaire.

SUMMARY:
Pseudoxanthoma elasticum (PXE) is a rare, autosomal recessive genetic disease characterized by progressive calcification and fragmentation of elastic fibers in connective tissues. PXE primarily affect the skin, retina and arterial walls. Given the age of onset and progression of the disease, the consequences of PXE affect a large number of patients of working age and are therefore likely to have an impact on their professional career and job retention.

To our knowledge, there are no studies on the occupational impact of PXE.

DETAILED DESCRIPTION:
This is an epidemiological, descriptive and analytical, cross-sectional, monocentric study, carried out by telephone questionnaire on the national cohort of the PXE Reference Center in the Dermatology Department of the Angers University Hospital.

Eligible subjects will be pre-selected by the study investigators on the basis of the medical file. A letter of information about the study will be sent to all the pre-selected eligible patients, with the exception of patients who have expressed an objection to the processing of their data for research purposes.

The investigators will contact eligible patients by telephone approximately 2 weeks after the mailing of the information letter. During this telephone call, the investigator will answer any questions the patient may have about the study and will collect the patient's non-objection to participate in the study and their responses to the questionnaire.

In the absence of a validated questionnaire to meet the objectives of the study, a questionnaire was created.

This questionnaire was tested in order to verify its feasibility and clarity. Medical data (age at diagnosis, age at referral to the Reference Centre, organ damage and clinical manifestations present at the time of the survey, treatments, etc.) will be collected from the medical file and the answers to the questionnaire will be collected by telephone on paper. Data will be collected in a coded manner. A correspondence list will be kept, under the responsibility of the principal investigator.

No follow-up of patients is planned by the study.

The results of this study should make it possible to provide new data on the impact of PXE on the career path and job retention of patients, as well as the medical reasons linked to it. It should also make it possible to improve knowledge on the experience of the consequences of PXE for patients in the workplace, as well as the actors and tools for job retention mobilised in these situations. All of these elements should make it possible to improve the prevention of the professional deintegration of PXE patients, in particular by setting up systematic and early management of patient-workers presenting a declared PXE.

ELIGIBILITY:
Inclusion Criteria:

* PXE
* Working age / Unemployed / Retired less than 2 years

Exclusion Criteria:

* Presence of one or more physical or psychological comorbidity likely to have an impact on the career path and job retention.
* Poor understanding of the french language
* Objection to participating in research

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: French PXE cohort (ClinicalTrials.gov Identifier: NCT01446380)
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Percentage of job loss due to PXE | At enrolment
  Percentage of patients whose employment was modified or discontinued due to PXE.

SECONDARY OUTCOMES:
Percentage of job loss due to the vascular impact | At enrolment
  Percentage of patients whose employment was modified or discontinued due to the vascular impact of PXE. Vascular impact will be assessed by their last Ankle Brachial Index measurement.
Percentage of job loss due to the visual impact | At enrolment
  Percentage of patients whose employment was modified or discontinued due to the visual impact of PXE. Visual impact will be assessed by their last Visual acuity measurement.
Percentage of job loss due to the skin impact | At enrolment
  Percentage of patients whose employment was modified or discontinued due to the skin impact of PXE. Skin impact will be assessed by the presence of skin damage due to PXE in the cervical and/or antecubital areas.

CONTACTS AND LOCATIONS:
Overall Officials: Denise JOLIVOT, MD, Study Chair — Clinical Research And Innovation Delegation Angers University Hospital
Locations (1):
- MARTIN Ludovic, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta MA, Gupta AK. Age and gender differences in the impact of psoriasis on quality of life. Int J Dermatol. 1995 Oct;34(10):700-3. doi: 10.1111/j.1365-4362.1995.tb04656.x. PMID 8537157
- [Result] Shimada BK, Pomozi V, Zoll J, Kuo S, Martin L, Le Saux O. ABCC6, Pyrophosphate and Ectopic Calcification: Therapeutic Solutions. Int J Mol Sci. 2021 Apr 27;22(9):4555. doi: 10.3390/ijms22094555. PMID 33925341
- [Result] Finger RP, Fenwick E, Marella M, Charbel Issa P, Scholl HP, Holz FG, Lamoureux EL. The relative impact of vision impairment and cardiovascular disease on quality of life: the example of pseudoxanthoma elasticum. Health Qual Life Outcomes. 2011 Dec 12;9:113. doi: 10.1186/1477-7525-9-113. PMID 22152229